CLINICAL TRIAL: NCT00793923
Title: A Prospective Study Comparing Ranibizumab Plus Dexamethasone Combination Therapy Versus Ranibizumab Monotherapy for Wet Age-related Macular Degeneration
Brief Title: A Prospective Study Comparing Ranibizumab Plus Dexamethasone Combination Therapy Versus Ranibizumab Monotherapy for Wet AMD
Acronym: Lucedex
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Subhransu K. Ray, M.D., Ph.D. (Other)
Collaborators: Bay Area Retina Associates (Other)
Responsible Party: Sponsor-Investigator, Subhransu K. Ray, M.D., Ph.D., Principal Investigator, Bay Area Retina Associates
Organization: Bay Area Retina Associates (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Lucedex
Record Dates: First submitted 2008-11-17; First posted 2008-11-19 (Estimated); Last update posted 2012-12-19 (Estimated); Status verified 2012-12

CONDITIONS: Exudative Age-Related Macular Degeneration
Keywords: Exudative Age Related Macular Degeneration
MeSH Terms: interventions — Ranibizumab; Dexamethasone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Combination Therapy (Experimental): Combination therapy (group 1): same day combination therapy with 0.05cc dose intravitreal dexamethasone injection (10mg/ml vial) and a single 0.5 mg intravitreal ranibizumab injection
  Interventions: Drug: ranibizumab and dexamethasone
- Monotherapy (Active Comparator): intravitreal injection of 0.5 mg ranibizumab
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: ranibizumab and dexamethasone — Combination therapy (group 1): same day combination therapy with 0.05cc dose intravitreal dexamethasone injection (10mg/ml vial) and a single 0.5 mg intravitreal ranibizumab injection
  Arms: Combination Therapy
Drug: Ranibizumab — intravitreal injection of 0.5 mg ranibizumab
  Arms: Monotherapy

SUMMARY:
The primary objective of this proposed research study is to evaluate the safety of intravitreal ranibizumab in combination with intravitreal dexamethasone in comparison to intravitreal ranibizumab alone in the treatment of wet ARMD. The addition of the broad spectrum anti-inflammatory activity of dexamethasone may augment the anti-VEGF activity of ranibizumab by amelioration of inflammation existing in the microenvironment of the choroidal neovascularization. While the anti-VEGF agents have proven to be very efficacious in the treatment of exudative ARMD, their narrow target and window of activity may limit their overall durability of action.

DETAILED DESCRIPTION:
A prospective, single masked comparative trial using either combination therapy (group 1): same day combination therapy with 0.05cc intravitreal dexamethasone injection (10mg/ml vial) and a single 0.5 mg intravitreal ranibizumab injection for four consecutive months will be compared to monotherapy (group 2): one intravitreal injection of 0.5 mg ranibizumab also given for four consecutive months. These treatments will then be followed by PRN treatment based on clinical exam, angiographic studies, and OCT evidence of residual subretinal fluid, CME, subretinal hemorrhage, or pigment epithelial detachment. Fluorescein angiography and fundus photography will be performed at baseline and at the 1, 3, 6, and 12 month follow-up visits. Only OCT testing will be performed at all follow-up visits. Both groups will be re-evaluated for safety at 12 and 24 months.

ELIGIBILITY:
Inclusion Criteria:

• Best Corrected Visual Acuity at 4 meters using ETDRS Charts between 20/32 and 20/400 (Snellen Equivalent) in the study eye with evidence of neovascular ARMD.

(Only one eye will be eligible for study. If both eyes are eligible, the one with the better visual acuity will be selected for treatment unless, based on medical reasons, the investigator deems the other eye to be more appropriate for treatment and study.)

* All lesion subtypes will be enrolled with the following criteria Predominantly and minimally classic: Angiographic lesion greater than 50% of the total lesion area Occult: Lesions must show recent activity progression with respect to vision, subretinal hemorrhage or subretinal fluid
* Signed informed consent
* Age greater than or equal to 50 years

Exclusion Criteria:

* Previous treatment for ARMD in the study eye
* Previous intravitreal drug delivery in the study eye
* Previous vitrectomy in the study eye
* Fibrosis or atrophy involving the center of the fovea in the study eye
* Neovascular membrane from any other concurrent retinal disease such as high myopia (SER > -8D), histoplasmosis or other ocular inflammatory disease.
* Known history of glaucoma and on more than one topical medication
* History of glaucoma filtering surgery in the study eye
* History of corneal transplant in the study eye
* Patients with active co-existing macular disease such as diabetic macular edema
* Active intraocular inflammation in the study eye
* History of allergy to fluorescein not amenable to treatment
* Pregnancy (positive pregnancy test) or lactation
* Premenopausal women not using adequate contraception. The following are considered effective means of contraception: surgical sterilization or use of oral contraceptives, barrier contraception with either a condom or diaphragm in conjunction with spermicidal gel, an IUD, or contraceptive hormone implant or patch.
* Any other condition that the investigator believes would pose a significant hazard to the subject if the investigational therapy were initiated
* Inability to comply with study or follow up procedures
* Participation in another simultaneous medical investigation or trial

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-01; Primary Completion 2012-01 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of ocular adverse events and visual acuity | 6 months and 12 months

SECONDARY OUTCOMES:
Total number of treatments required | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Subhransu K Ray, M.D., Ph.D., Principal Investigator — Bay Area Retina Associates
Locations (1):
- Bay Area Retina Associates, Walnut Creek, California, United States